CLINICAL TRIAL: NCT03309072
Title: Investigating Accelerated Learning and Memory in Healthy Subjects Using a Face Name Memory Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-96
Record Dates: First submitted 2017-10-07; First posted 2017-10-13 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Healthy Adults
Keywords: transcranial Direct Current Stimulation (tDCS); accelerated learning; memory
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: (1) active tDCS with Face Name associate memory task (2) sham tDCS with Face Name associate memory task
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active tDCS (Experimental): active tDCS with Face Name associate Memory task
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): sham tDCS with Face Name associate Memory task
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — active tDCS
  Arms: active tDCS
Device: sham tDCS — sham tDCS
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to investigate whether we can accelerate learning and improve associative memory performance in healthy subjects by applying transcranial Direct Current Stimulation (tDCS) during a Face Name memory task.

DETAILED DESCRIPTION:
Associative memory refers to remembering the association between two items, such as a face and a name or a word in English and the same word in another language. It is not only important for learning, but it is also one of the first aspects of memory performance that is impacted by aging and by Alzheimer׳s disease. For decades, neuroscientists have investigated associative learning and memory and ways to accelerate and enhance associative learning and memory.

Transcranial Direct Current stimulation (tDCS) is a non-invasive and painless electrical stimulation technique that has demonstrated to accelerate learning and improve memory in some studies. To investigate whether we can accelerate learning and improve associative memory using tDCS, we will compare the performance in a Face Name Associate memory task from 2 groups. The first group will get active tDCS during the study phase of the Face Name Memory task, whereas the second group will get sham tDCS during the study phase of the task.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Native English Speaker

Exclusion Criteria:

* History of severe head injuries, epileptic insults, or heart disease.
* Severe psychiatric disorders and severe untreated medical problems.
* Contraindications for tDCS (pregnant women, implanted devices)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas of Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Age between 18 and 35
  2. Currently not using any medication
  3. Native English speaker
  4. Capable of understanding and signing an informed consent
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.67 (2.5) | 20.6 (3.9) | 20.13 (3.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 4 | 10
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Beck Depression Inventory Scale [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI, BDI-1A, BDI-II), created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  The Beck Depression Inventory uses the following scale to assess patients: 0 - 13: Minimal depression, 14 - 19: Mild depression, 20 - 28: Moderate depression, 29 - 63: Severe depression
  Min score: 0; Max Score: 63; The higher the score the more mood
  units on a scale | 5.20 (3.61) | 3.47 (3.62) | 4.33 (3.66)
Beck Anxiety Inventory Scale [Mean (Standard Deviation); unit: units on a scale] — The Beck Anxiety Inventory (BAI), created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.
  The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs[4] are:
  0-7: minimal anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
  units on a scale | 4.53 (3.38) | 2.67 (2.85) | 3.60 (3.21)
Mini Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
  Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
  units on a scale | 28.9 (0.88) | 28.5 (1.51) | 28.7 (1.24)
Profile of Mood States- Mood Disturbance [Mean (Standard Deviation); unit: units on a scale] — The Profile of Mood States (POMS) is a psychological rating scale used to access transient, distinct mood states. The total score is reported.
  The higher the score the more people are sensitive to mood swings.
  Min score 0 - Max score is 148.
  units on a scale | 10.27 (23.2) | 1.47 (11.33) | 4.4 (18.9)

OUTCOME MEASURES:

1. Primary Outcome: Associative Memory Assessed by a Face Name Associate Memory Experiment
Description: All participants performed a face memory task .The face stimuli consisted of 120 grayscale pictures of human faces. Only faces with a neutral expression facing forward were selected. Half of the faces were male, and the other half were female. The face-name association memory task was divided into (1) an encoding phase, (2) a consolidation phase, and (3) a retrieval phase. During the encoding phase, participants studied 60 successively presented face-name pairs and were instructed to assess their gender to keep them focused to the task. The encoding phase was followed by a consolidation phase where participants were instructed to "sit still, relax, and think about nothing in particular" for 10 minutes, During the retrieval phase, participants were presented with 60 old and 60 new faces and were instructed to assess whether they have seen this face during the encoding phase.
  The outcome was the percent of Correct Name to Face Matches
Time Frame: Associate Memory is assessed after a 10 minutes break following the study phase
Measure: Mean (Standard Deviation); unit: Percent of Correct Name to Face Matches
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 15
Percent of Correct Name to Face Matches | 44.22 (11.54) | 35.44 (12.04)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Other — To compare the old and new faces' hit rate, we calculated the true positive rate (TPR: the proportion of positives that are correctly identified as such). A repeated measures ANOVA was conducted with the TPR for both old and new faces as within-subjects variable and group (active vs sham) as between-subjects variable; p < .049, ANOVA; Mean Difference (Net) = 10.66 — Difference between active tDCS and sham tDCS

ADVERSE EVENTS:
Time Frame: 1 week
Description: At the end of the stimulation procedure, participants complete an exit questionnaire on which they can report side-effects from the study.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol: Protocol 17-96 (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03309072/Prot_001.pdf